CLINICAL TRIAL: NCT03406234
Title: Observational Study on the Risk Factors for Health in a Chinese Population
Brief Title: Observational Study on a Chinese Population
Status: Completed | Type: Observational
Sponsor: Shenzhen Center for Chronic Disease Control (Other)
Responsible Party: Principal Investigator, Zhou Ji-Chang, Director of Molecular Biology Laboratory, Shenzhen Center for Chronic Disease Control
Other Study IDs: QLS2013
Record Dates: First submitted 2018-01-08; First posted 2018-01-23 (Actual); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Metabolic Disease; Nutrition Disorders; Genetic Predisposition to Disease
MeSH Terms: conditions — Metabolic Diseases; Nutrition Disorders; Genetic Predisposition to Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- A group of participants
  Interventions: Other: No intervention.

INTERVENTIONS:
Other: No intervention. — Cross-sectional observation without interventions.

SUMMARY:
An observational study was conducted in a health examination center to distinguish risk factors for health in a randomly recruited volunteers of Chinese population.

ELIGIBILITY:
Inclusion Criteria:

* Han population, living in Shenzhen City for > 2 y, not in pregnancy, without hepatic diseases and renal diseases

Exclusion Criteria:

* caught by organic diseases

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Both males and females were included.
Sampling Method: Probability Sample
Enrollment: 2650 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2013-12-31 (Actual); Study Completion 2013-12-31 (Actual)

PRIMARY OUTCOMES:
Circulating 25OHD concentration. | Jan., 2014 - May., 2015

SECONDARY OUTCOMES:
Body mass index | Jan.-Dec., 2013
Plasma glucose | Jan.-Dec., 2013
DNA polymorphisms | Jan., 2014 - Dec., 2017
Plasma lipids | Jan.-Dec., 2013
Blood pressure | Jan.-Dec., 2013

CONTACTS AND LOCATIONS:
Locations (1):
- Shenzhen Center for Chronic Disease Control, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chen J, Yun C, He Y, Piao J, Yang L, Yang X. Vitamin D status among the elderly Chinese population: a cross-sectional analysis of the 2010-2013 China national nutrition and health survey (CNNHS). Nutr J. 2017 Jan 14;16(1):3. doi: 10.1186/s12937-016-0224-3. PMID 28088200
- [Result] Santos BR, Mascarenhas LP, Boguszewski MC, Spritzer PM. Variations in the vitamin D-binding protein (DBP) gene are related to lower 25-hydroxyvitamin D levels in healthy girls: a cross-sectional study. Horm Res Paediatr. 2013;79:162-8. doi: 10.1159/000348847. Epub 2013 Mar 20. PMID 23548751
- [Result] Gozdzik A, Zhu J, Wong BY, Fu L, Cole DE, Parra EJ. Association of vitamin D binding protein (VDBP) polymorphisms and serum 25(OH)D concentrations in a sample of young Canadian adults of different ancestry. J Steroid Biochem Mol Biol. 2011 Nov;127(3-5):405-12. doi: 10.1016/j.jsbmb.2011.05.009. Epub 2011 Jun 12. PMID 21684333
- [Derived] Zhou JC, Zhu Y, Gong C, Liang X, Zhou X, Xu Y, Lyu D, Mo J, Xu J, Song J, Che X, Sun S, Huang C, Liu XL. The GC2 haplotype of the vitamin D binding protein is a risk factor for a low plasma 25-hydroxyvitamin D concentration in a Han Chinese population. Nutr Metab (Lond). 2019 Jan 14;16:5. doi: 10.1186/s12986-019-0332-0. eCollection 2019. PMID 30651747